CLINICAL TRIAL: NCT05668325
Title: INVESTIGATION OF THE EFFECT OF HOME BASED MINI TRAMBOLINE EXERCISE PROGRAM ON DIABETIC FOOT CARE BEHAVIOR AND DIABETIC POLYNEUROPATHY
Brief Title: The Effect of Mini Trampoline Exercise Program on Diabetic Foot Care Behavior and Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Buket DAŞTAN, Lecturer phd, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCS16956037
Record Dates: First submitted 2022-12-10; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Polyneuropathy; Diabetic Foot; Type 2 Diabetes
Keywords: Behavior; Diabetic foot; Diabetic polyneuropathy; Exercise; Range of motion
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot; Diabetes Mellitus, Type 2; Behavior; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The number of samples was determined by using the G*Power 3.1.9.6 program with a 95% confidence interval of 0.05 error rate, a study in which the effects of the mini trampoline exercise program performed with diabetic polyneuropathy patients on foot mobility and foot sensation in the literature were evaluated, with a power of 80% and an effect size of 0.90. calculated. As a result of the statistical analysis, it was found that a total of 28 patients, 14 in the mini trampoline exercise group and 14 in the control group, should be included in the study. Considering that if the sample size increases, the standard error will decrease and the working power will increase, each group was increased by 43% and a total of 40 patients were included in the study, 20 patients for each group.
Who Masked: Participant
Masking Description: The block randomization method was applied. The coin flip method was used to determine the exercise and control groups, and the exercise group was determined as A and the control group B. In our study, in which octal blocking was performed with four A and four B blocks in each block, the possible number of blocks was calculated as 70. Five numbers between 1 and 70 were generated (for 40 people, it is enough to choose five random blocks) using the "in randomear" command in Excel, and the numbers 27, 11, 13, 18, 51 were obtained. Patients were randomized according to the blocks corresponding to these numbers. In addition, in the "post-hoc" power analysis performed at the end of the study, the power of the study was determined to be 85%, and this result showed that the sample size of the study was sufficient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini trampoline exercise group (Experimental): "Structured Patient Information Form" and "Foot care behavior scale", "5.07/10 g Semmes-Weinstein Monofilament", "128 Hz Manual Electronic Tunnel" and "Goniometer" were applied to the patients as a pre-test and recorded in the patient registry. related forms. Afterwards, diabetic foot care information was given to the patients and "Diabetic Foot Care Information Brochure" was given. Afterwards, the patients were visited for a total of 24 times a week, three days a week for eight weeks. At the first visit, the patients were informed about the exercise program and then the "Home-based Mini Trampoline Exercise Information Brochure" was given to the patients. The patients were given an exercise program three times a week, a total of 24 times for eight weeks. In addition, the "Foot Monitoring Form" was applied to the patients once a week. Apart from the "Structured Patient Information Form", other data collection tools were applied to this patient group as a post-test.
  Interventions: Other: Mini trampoline exercise group
- Control group (Experimental): Data collection tools were applied to this group of patients before the study. Diabetic foot care information was given and "Diabetic Foot Care Information Brochure" was given. A total of eight home visits were made for eight weeks, once a week, and the "Foot Monitoring Form" was applied. At the end of eight weeks, all data collection tools except the "Structured Patient Information Form" were applied again.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Mini trampoline exercise group — In this study, patients performed a 30-45 minute mini-trampoline exercise program 3 times a week for eight weeks (two months) under the supervision of the investigator.
  Arms: Mini trampoline exercise group
Other: Control group — In this study, patients were visited at home once a week for eight weeks and their feet were checked.
  Arms: Control group

SUMMARY:
This study was planned to examine the effect of home-based mini trampoline exercise program on diabetic foot care behavior and diabetic polyneuropathy in Type 2 diabetes patients.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a rapidly increasing metabolic disease in the world. It is stated that the incidence of DM, one of the most important public health problems, is increasing much faster than in the past, and it is estimated that approximately 592 million people will be affected worldwide by 2035. Diabetic foot; represents a range of complications caused by a combination of neuropathy and varying degrees of vascular disease in diabetic patients, including lower extremity infection, ulcer formation, and/or deep tissue damage. Diabetic foot is the cause of approximately 75-85% of all lower extremity amputations. Diabetic foot is also the leading cause of non-traumatic lower extremity amputations worldwide. Diabetic polyneuropathy is a peripheral neuropathy characterized by symmetrical sensory symptoms such as numbness, paresthesia, pain and muscle weakness predominantly in the distal parts of the arms and legs. Diabetic neuropathy is one of the most common complications of diabetes and its lifetime prevalence exceeds 50%, especially in Type 2 diabetes patients.

Prevention of diabetic foot is possible by adopting healthy foot care behaviors and applying examination methods that evaluate foot health. It is reported that it is important to evaluate autonomic neuropathy symptoms (skin dryness, hydration, color) and motor neuropathy symptoms (weakening of the inner foot muscles, foot deformities) in the foot examination of the patients. In addition, it is stated that the diabetic polyneuropathy symptom of the patients should be measured using the "semmes-weinstein 10 g monofilament" protective sense, the "128 Hz tuning fork" vibration perception and the "goniometer" to measure the ankle and 1st metatarsophalangeal joint (MTPJ) mobility. There are important findings on the effectiveness of regular physical activity in the prevention of primary and secondary development of diabetes and diabetic foot. Today, supervised exercise programs in the home environment are supported to ensure the continuity of exercise of the patients and the demand for exercises that can be applied at home is increasing. Exercise programs performed at home under the supervision of a professional provide a structured program, increase self-motivation through feedback, and encourage participants to exercise. In the literature, it is stated that supervised foot exercises, together with a health-promoting program, effectively reduce the symptoms of diabetic neuropathy, improve vibration perception and joint mobility of the foot and ankle, redistribute pressure during walking, and increase foot strength and function. These positive effects also reduce the risk factors for the development of foot ulcers in diabetes.

While there are guidelines and studies on exercise practice in diabetes management in Turkey, there are gaps in the literature and practices regarding diabetic foot care behaviors and foot exercises in diabetic polyneuropathy. Therefore, it would be beneficial to explore alternative, easy exercises to manage diabetes and prevent/delay diabetic foot complications and promote care. In this study, it was aimed to examine the effect of home-based mini trampoline exercise program on foot care behaviors and diabetic polyneuropathy in Type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type 2 diabetes and diabetic polyneuropathy for at least one year,
* Having a body mass index between 18-30 kg/m2,
* Being literate,
* Being residing in XXXX province,
* Was determined as agreeing to participate in the study.

Exclusion Criteria:

* Having a history of malignancy,
* Myocardial infarction, stroke, liver failure/renal failure, foot/leg amputation,
* Current or previous foot ulcer,
* History of surgery on the knee, ankle or hip, major vascular complications and/or severe retinopathy,
* Dementia or not being able to give consistent information,
* Doing regular exercise such as walking, running or foot exercise,
* Receiving physiotherapy at any time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | 8 week.
  This form included 15 questions to determine the sociodemographic characteristics of the patients (age, BMI, gender, marital status, education level, occupation, income perception level, smoking status) and disease-related characteristics.
  The mini-trampoline exercise group was administered to the patients twice before the study and at the end of the 8th week.
Foot Care Behavior Scale | 8 week.
  It was created by Borges in 2007 with the aim of improving foot self-care behaviors in diabetes. The one-dimensional scale consists of 15 items; The items consist of a five-point Likert scale. The scale score is calculated as the lowest 15 and the highest 75 points. An increase in the score obtained from the scale indicates that the patient's self-care behaviors are better.
  The mini-trampoline exercise group was administered to the patients twice before the study and at the end of the 8th week.
Foot Tracking Form | 8 week.
  It was created by the researcher to use in the foot follow-up of patients by scanning the literature on diabetic foot. in form; "Washing, drying, moisturizing, foot control, socks change, shoe change, shoe control, foot positioning and nail cutting", which includes the foot care behaviors of the patients, took place.
  It was applied to the patients once every week, a total of 8 times.
Home Based Mini Trampoline Exercise Tracking Form | 8 week.
  The home-based mini trampoline exercise monitoring form was created by the researcher to be used in the follow-up of the patients' home-based mini trampoline exercise program by scanning the literature on mini trampoline exercises. In form; each patient-specific exercise day, exercise time, exercise duration, exercise break time, and post-exercise foot control were included.
  It was applied to the patients once every week, a total of 8 times.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayburt University, Bayburt, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I'll decide later